CLINICAL TRIAL: NCT04863365
Title: A Multi-center, Randomized, Placebo-controlled, Double-blind, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of PHP-201 in Patients With Primary Open-angle Glaucoma or Ocular Hypertension
Brief Title: A Study of Efficacy and Safety of PHP-201 in Patients With Primary Open Angle Glaucoma or Ocular Hypertension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: pH Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHP-201-S301
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-04

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Primary Open-angle Glaucoma; ROCK inhibitor
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — sovesudil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo treatment (Placebo Comparator): A matching placebo ophthalmic solution, TID
  Interventions: Drug: Placebo ophthalmic solution
- PHP-201 treatment (Experimental): PHP-201 0.5% ophthalmic solution, TID
  Interventions: Drug: PHP-201 ophthalmic solution

INTERVENTIONS:
Drug: Placebo ophthalmic solution — A matching placebo ophthalmic solution, 3 drops daily, 28 days
  Other Names: Matching placebo
  Arms: Placebo treatment
Drug: PHP-201 ophthalmic solution — PHP-201 0.5% ophthalmic solution, 3 drops daily, 28 days
  Other Names: Sovesudil
  Arms: PHP-201 treatment

SUMMARY:
This is a phase 3 study to confirm the efficacy in reduction of intraocular pressure and safety of PHP-201 ophthalmic solution in patients with primary open-angle glaucoma or ocular hypertension.

DETAILED DESCRIPTION:
As a selective ROCK inhibitor, PHP-201 is designed to alleviate the side effects, which are the disadvantages of existing intraocular pressure reducing agents, while exhibiting sufficient intraocular pressure-lowering effect in glaucoma patients. This clinical trial aims to provide a new therapeutic option by evaluating the efficacy and safety of PHP-201 0.5% in patients with primary open-angle glaucoma or ocular hypertension who require intraocular pressure reduction therapy.

ELIGIBILITY:
Subject Inclusion Criteria:

1. The age of 19 years or older
2. Diagnosis of open-angle glaucoma (POAG) or ocular hypertension (OH)
3. Intraocular Pressure(IOP) ≤ 35mmHg at both eye and IOP ≥ 22mmHg at either eye
4. Shaffer's grading > 2
5. Best-corrected visual acuity in both eye equivalent to 0.2logMar
6. Able and willing to give signed informed consent

Subject Exclusion Criteria:

1. Central corneal thickness <500㎛ or >600㎛
2. Medical history of following

   * Closed-angle glaucoma, pigment dispersion syndrome, pseudoexfoliation, narrow-angle glaucoma
   * Advanced glaucomatous loss; mean deviation (MD) < -12dB
   * Moderate to severe inflammatory/infectious disease in either eye
   * Advanced retinopathy
   * Surgical or laser therapy for glaucoma treatment
3. Have confirmed the following at the screening visit

   * SBP ≥ 180mmHg or DBP ≥ 110mmHg
   * HbA1c > 9.0%
   * CrCl < 30mL/min
   * AST or ALT ≥ 3 X ULN
   * Unstable angina, myocardial infarction, transient ischemic attack, cerebral stroke, coronary artery bypass graft, or coronary angioplasty within 24 weeks
   * History of malignant tumor with 5 years
   * History of the causative disease that may cause secondary glaucoma, including a history of steroid administration for more than 4 weeks
4. Conditions need to wear contact lenses during the study
5. Known hypersensitivity to any component of the investigational product
6. Who has administered topical/systemic drugs that may affect the study within a certain period prior to eligibility check or are expected to need administration during the study duration

   * Prostaglandin analogues: 5 weeks
   * β-blockers: 4 weeks
   * ROCK inhibitors: 4 weeks
   * α/β-adrenergic agonists: 2 weeks
   * Muscarinic agonists: 1 week
   * Carbonic anhydrase inhibitors: 1 week
   * Systemic corticosteroids: 4 weeks
7. Pregnant or breast-feeding
8. Who disagreed with the use of the methods of proper contraception during the study duration
9. Administration or use of other investigational drugs/devices prior to the screening visit within its 5 half-lives or 30 days, whichever is longer
10. Unsuitable for participation in the study according to the judgment of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure | 4 weeks
  Mean IOP change from baseline

SECONDARY OUTCOMES:
Diurnal intraocular pressure | 4 weeks
  Mean of diurnal IOP change from baseline

OTHER OUTCOMES:
Treatment-emergent adverse event | up to 6 weeks
  Safety assessed by number of participants experienced treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Younyoung Hwang, Study Director — pH Pharma
Locations (1):
- Seoul National University Hopsital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No